CLINICAL TRIAL: NCT05642767
Title: Molecular Detection Of Efflux Pump and Virulence Factors Genes in Pseudomonas Aeruginosa
Acronym: Pseudomonas
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Noha Saber Shafik, lecturer of Medical Microbiology and Immunology, faculty of medicine, Sohag University
Other Study IDs: Soh-Med-22-11-18
Record Dates: First submitted 2022-11-19; First posted 2022-12-08 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Pseudomonas Aeruginosa
Keywords: Efflux genes, Pseudomonas , virulence, PCR
MeSH Terms: conditions — Pseudomonas Infections; Pathologic Complete Response | interventions — Staining and Labeling

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Samples (pus, urine, blood, sputum, ear discharge) will be collected from different departments at sohag university hospital.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with pseudomonas aeruginosa infections: All patients suffer from infections that can be caused by pseudomonas aeruginosa.
  Clinical Data will be obtained as:
  * Data about clinical manifestations including fever, expectoration, pus from wounds, urinary symptoms, symptoms of upper respiratory tract infections, and symptoms of otitis externa.
  * Samples will be cultured on cetrimide agar.
  * Antibiotic sensitivity testing will be done by disc diffusion method according to CLSI.
  * Molecular detection to efflux genes and some virulence genes by PCR.
  Interventions: Diagnostic Test: culture on cetrimide agar; Diagnostic Test: Staining with Gram stain; Diagnostic Test: Antibiotic sensitivity testing; Diagnostic Test: Molecular detection to efflux genes and some virulence genes
- Patients with infections other than pseudomonas aeruginosa: * Data about clinical manifestations including fever, expectoration, pus from wounds, urinary symptoms, symptoms of upper respiratory tract infections, and symptoms of otitis externa.
  * Samples will be cultured on different culture media and automated identification by Vitek system.
  Interventions: Diagnostic Test: culture on cetrimide agar; Diagnostic Test: Staining with Gram stain; Diagnostic Test: Antibiotic sensitivity testing

INTERVENTIONS:
Diagnostic Test: culture on cetrimide agar — Samples will be inoculated on cetrimide agar using the plating out technique.
Diagnostic Test: Staining with Gram stain — colonies on cetrimide agar will be spread on glass slide and stained by gram stain
Diagnostic Test: Antibiotic sensitivity testing — Antibiotic sensitivity testing will be done by disc diffusion method according to CLSI
Diagnostic Test: Molecular detection to efflux genes and some virulence genes — Molecular detection to efflux genes and some virulence genes by conventional PCR
  Groups: Patients with pseudomonas aeruginosa infections

SUMMARY:
Pseudomonas aeruginosa (PA) is a ubiquitous aerobic, non-fermentative Gram-negative rod that is widely associated with nosocomial pneumonia and can lead to severe illness with poor outcomes, particularly in critically ill people due to the ability of some strains to cause lung epithelial injury and spread into the circulation. 2 In the intensive care unit, PA infection is ranked among the top five causes of the bloodstream, pulmonary, surgical site, urinary tract, and soft tissue infections.

DETAILED DESCRIPTION:
The pathogenesis of PA infections is multifactorial, and it is frequently complicated by the bacteria's intrinsic resistance to some antimicrobial agents such as sulfonamides, tetracyclines, and trimethoprim, as well as its ability to acquire or quickly develop resistance to major classes of antibiotics such as aminoglycosides, quinolones, B-lactams, and polymyxins (Bassetti et al., 2018).

The efflux systems, which mediate the expulsion of antibiotics out of the cell shortly after entry, the production of enzymes to inactivate antibiotics, and the decrease in permeability across the cell wall are some mechanisms used by PA to develop antimicrobial resistance (Meletis & Bagkeri, 2013).

PA possesses a large number of virulence factors that play a significant role in pathogenesis and the determination of infection severity. These virulence factors act alone or in synergy with each other to cause tissue damage, necrosis, and cell death. Among the virulence factors of PA, the major determinants of virulence are the type III secretion system (T3SS) and quorum sensing (cell-to-cell signaling system). The T3SS is a needle-like complex, also known as the injectisome, that enables a bacterium to deliver different effector proteins such as ExoS, ExoT, ExoU, and ExoY across the membrane into a host cell, altering host cell functions and increasing bacterial survival rates ( Horna G and, Ruiz J, 2021). In this study, we aimed to evaluate the prevalence of antibiotic resistance caused by the presence of Efflux genes and some virulence factors in Pseudomonas aeruginosa from clinical isolates.

ELIGIBILITY:
Inclusion Criteria:

* All patients suffering from infections that can be caused by pseudomonas aeruginosa

Exclusion Criteria:

* Samples diagnosed to have organisms other than pseudomonas aeruginosa.

Ages: 4 Weeks to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will be carried out on all patients suffering from infections that can be caused by pseudomonas aeruginosa.
  Samples (pus, urine, blood, sputum, ear discharge) will be collected from different departments at sohag university hospital.
  Clinical Data will be obtained as:
  - Data about clinical manifestations including fever, expectoration, pus from wounds, urinary symptoms, symptoms of upper respiratory tract infections, and symptoms of otitis externa.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Isolation and identification of pseudomonas aeruginosa using culture and automated system techniques | 1 December 2022 to 1 February 2023
  identification of pseudomonas aeruginosa in different clinical samples collected from Sohag University hospital using different laboratory techniques as culture on citramide agar, Staining with Gram, biochemical reactions such as Oxidase test, sugar fermentation test, and automated identification using vitek2 system
Identification of recent antibiotic sensitivity pattern using Modified Kerby -Disc Diffusion method | 1 December 2022 to 1 February 2023
  Determination of recent antibiotic sensitivity pattern using different antibiotics by disc diffusion method by spreading the inoculum in pitry dish containing Muller Hinton Agar, then different discs containing antibiotics are placed at a distance of 1.5 cm, then incubated at 37 co for 24 hrs. The diameter of the zone of inhibition is measured to determine MIC for each antibiotic according to the guidelines of CSLI 2022.
Molecular Identification of some virulence factors and efflux genes using PCR | 1 February 2023 to 30 March 2023
  Molecular detection of some virulence factors and efflux genes using specific primers by conventional PCR. primers of the following genes will be used as exoS,exoU, toxA, mex A, mex B. Extraction of DNA will be done first, followed by amplification technique using the thermal cycler. Detection of amplified DNA will be done using Agrose gel electrophoresis stained with ethidium bromide.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed H Alrawy, Study Chair — Faculty of medicine, Sohag university; Ebtisam M Gad, Study Chair — Faculty Of Medicine, Sohag university
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://doi.org/10.5772/55616